CLINICAL TRIAL: NCT02515370
Title: Using Enhanced Peer Group Strategies to Support Prevention of Mother to Child HIV Transmission (PMTCT) Option B+ in Uganda
Brief Title: Friends for Life Circles for Option B Plus
Acronym: FLCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MU-JHU CARE (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Philippa Musoke, MBChB, PhD, Site Leader, MU-JHU CARE
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Musoke-R01-080476-Option B+
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: Option B plus; HIV infected women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Friends for Life Circles (FLC) (Experimental): The intervention will include formation of peer support groups of eight to ten women in the community with incorporation of income generating activities to improve maternal adherence to clinic appointments and life long antiretroviral therapy
  Interventions: Other: Friends for Life Circles (FLCs).
- Standard of Care (SOC) (No Intervention): Normal standard of care and follow up. The standard care provided in the clinic will be provided for the control arem

INTERVENTIONS:
Other: Friends for Life Circles (FLCs). — The intervention 'Friends for Life Circles" (FLCs) will build dynamic peer group support in the community aimed at supporting maternal adherence to appointment keeping and taking lifetime antiretroviral drugs
  Arms: Friends for Life Circles (FLC)

SUMMARY:
The main goal of the study is to support HIV-infected pregnant women initiated on PMTCT Option B+ during antenatal to adhere to lifelong ART and postpartum care visits through an enhanced group peer support intervention called "friends for life circles".

DETAILED DESCRIPTION:
The overall goal of this implementation research is to improve retention in care and adherence to ART to 2 years postpartum among HIV infected women in urban and rural Uganda choosing PMTCT Option B+. Formative research will first be conducted to assess knowledge and attitudes regarding Option B+ and lifelong ART among PMTCT clients, community members and health workers. The formative research will inform the design of the group peer support intervention. Interventional research will then be conducted randomizing 540 women to either enhanced group peer support with income generating activities called the Friends for Life Circle (FLC) or MOH standard of care counselling with follow-up to 2 years postpartum. Primary outcomes will include retention in health care, ARV adherence and viral suppression at 6 weeks and 24 months postpartum. Secondary outcomes will include participants' health and economic outcomes.

ELIGIBILITY:
Inclusion criteria

* Age >18 years
* Documentation of pregnancy through clinical assessment or pregnancy test
* Documentation of confirmed HIV-positive sero-status at the time of screening
* Accepting to receive option B+ for PMTCT
* Providing written informed consent to participate in the randomized trial.
* Agreeing to come the study clinic for scheduled appointments
* Agreeing to be home visited as needed to ensure follow up
* Residing within a 20 km radius around the study clinic
* Not planning to move out of the catchment area within the next 2 years

Exclusion criteria

- Social and other circumstances that may prevent the mother from coming back for follow up

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 540 (Actual)
Dates: Start 2016-05; Primary Completion 2019-05 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Retention | 2 years
  in care will be measured as 1 minus proportion of women lost to follow-up at 24 months postpartum
Adherence to Option B+ ARV drugs | 2 years
  compare maternal antiretroviral drug adherence using self-report, viral load in blood at delivery, 6 weeks, 6 and 24 months postpartum among all HIV-infected pregnant women participating in the study.

SECONDARY OUTCOMES:
Infant HIV Free survival | 2 years
  also compare infant HIV-free survival at 6 weeks and 18 months among women randomized to the enhanced community-based intervention (FLC) versus the MOH SOC. Infants born to HIV-infected mothers are tested routinely at 6 weeks of
  age for HIV DNA by PCR and at 18 months of age by rapid HIV antibody test as part of the national Early Infant HIV Diagnosis program which is standard of care in every government health unit offering postnatal care in Uganda
Assessing success and sustainability of FLCs group support activities and IGAs | 2 years
  Each FLC will be assessed to see which groups were most successful in developing specific IGAs. The evaluation will be focus on the ability of FLCs to effectively generate income, participant attendance to the circles' IGA-related activities, key skills gained by participants in the circles and the percent increase or decrease in personal and household income

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Musoke, MD PhD, Principal Investigator — MU-JHU CARE
Locations (1):
- MUJHU Research Collaboration, Kampala, Uganda

REFERENCES:
- [Derived] Amone A, Gabagaya G, Wavamunno P, Rukundo G, Namale-Matovu J, Malamba SS, Lubega I, Homsy J, King R, Nakabiito C, Namukwaya Z, Fowler MG, Musoke P. Enhanced peer-group strategies to support the prevention of mother-to-child HIV transmission leads to increased retention in care in Uganda: A randomized controlled trial. PLoS One. 2024 Apr 19;19(4):e0297652. doi: 10.1371/journal.pone.0297652. eCollection 2024. PMID 38640123
- [Derived] Gabagaya G, Rukundo G, Amone A, Wavamunno P, Namale-Matovu J, Lubega I, Nakabiito C, Namukwaya Z, Nolan M, Malamba SS, King R, Homsy J, Fowler MG, Musoke P. Prevalence of undetectable and suppressed viral load in HIV-infected pregnant women initiating Option B+ in Uganda: an observational study nested within a randomized controlled trial. BMC Infect Dis. 2021 Sep 4;21(1):907. doi: 10.1186/s12879-021-06608-4. PMID 34481464